CLINICAL TRIAL: NCT06730672
Title: Efficacy and Safety of Voronib Combined With Everolimus After Immunotherapy Failure in Advanced Renal Carcinoma
Brief Title: An Exploratory Study on the Failure of Immunotherapy With Voronib Combined With Everolimus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-659-01
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Renal Cell Carcinoma Stage I
Keywords: Renal Cell Carcinoma; Failure in immune checkpoint inhibitors renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volonib combined with Everolimus Formation (Experimental): Volonib 200mg once daily and Everolimus 5mg once daily
  Interventions: Drug: Volonib combined with Everolimus Formation

INTERVENTIONS:
Drug: Volonib combined with Everolimus Formation — Volonib 200mg once daily and Everolimus 5mg once daily
  Other Names: Single-arm

SUMMARY:
This single-arm exploratory study included patients with renal clear cell carcinoma who had previously received one type of immunotherapy and failed. The specific regimen was Voronib 200mg PO.QD combined with everolimus 5mg QD. 80 patients were planned to continue treatment until PD, toxicity became intolerable, patient withdrawal was informed, or medication had to be discontinued. Collect patient medication information and disease efficacy evaluation, adverse reactions. In this study, blood samples were collected 0-4 weeks before treatment, 2 months, 4 months, 6 months, 8 months of drug treatment, and at the time of PD progression for ctDNA detection.

DETAILED DESCRIPTION:
The participant must have received no more than two kinds of tyrosine kinase inhibitors (TKIs) medications (excluding mTOR inhibitors) and one type of immune checkpoint inhibitor treatment, with treatment failure in systemic antitumor therapy. Additionally, the participant must have completed the last systemic antitumor treatment ( chemotherapy,radiotherapy, targeted therapy, biological therapy, or endocrine therapy) at least 3 weeks prior, or at least 5 half-lives since the last systemic antitumor treatment. Furthermore, any treatment-related toxicities must have resolved to meet the laboratory test requirements for this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Clear cell carcinoma of the kidney is confirmed by pathology (histology or cytology);
2. Have received systemic anti-tumor therapy with no more than 2 targeted drugs (excluding mTOR inhibitors) and 1 immune checkpoint inhibitor and failed treatment;
3. Not less than 3 weeks after receiving the last systemic anti-tumor therapy (chemotherapy, radiotherapy, targeted therapy, biotherapy or endocrine therapy), Or not less than 5 half-lives since the last systemic antitumor treatment; And treatment-related toxicity was recovered to meet the laboratory test requirements for this study;
4. ECOG score ≤ 1;
5. Over 18 years old, and less than or equal to 75 years old; a life expectancy of more than 12 weeks
6. According to RECIST 1.1 criteria: at least one measurable lesion;
7. Organ function levels must meet the following requirements:

   Bone marrow: blood test results must show hemoglobin ≥ 80 g/L, platelets ≥ 90 x 10^9/L, absolute neutrophil count ≥ 1.5 x 10^9/L; Liver: serum bilirubin ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (if there is liver metastasis, AST and ALT ≤ 5 times the upper limit of normal are allowed); Serum creatinine < 1.5 times the upper limit of normal; Urinary protein ≤ 2+, if urinary protein > 2+, a 24-hour urine protein test must be collected with a total amount ≤ 2 grams; Well-controlled hypertensive patients; Echocardiogram shows left ventricular ejection fraction greater than 40%;
8. For women of childbearing potential, the serum pregnancy test must be negative within 7 days prior to randomization;
9. All enrolled subjects (regardless of gender) must use effective barrier contraceptive methods throughout the treatment period and for 4 weeks after treatment ends;
10. Subjects must have the ability to understand and voluntarily sign the informed consent form, and the signing of the informed consent must occur prior to any study procedure.

Exclusion Criteria:

1. Previously only received single-drug targeted drug therapy against VEGF/VEGFR or mTOR；
2. Subjects currently receiving antitumor therapy (e.g., chemotherapy, radiation therapy, immunotherapy, biotherapy, hormone therapy, surgery, and/or tumor embolization, but excluding local radiation therapy for bone metastases) may be enrolled if they have a half-life of 5 years after the end of drug therapy；
3. Progression after previous mTOR therapy (monotherapy or combination)；
4. Conditions of the subjects' organ systems:

   Presence of significant pleural effusion or ascites with clinical symptoms requiring symptomatic treatment; brain metastases, or epidural metastases;
5. Subjects who have had other malignancies within the past 5 years (excluding non-melanoma skin cancer, cervical carcinoma in situ, or successfully treated basal cell carcinoma or squamous cell carcinoma);
6. Any uncontrolled clinical issues, including but not limited to, persistent or active infections, uncontrolled diabetes, decompensated liver cirrhosis;
7. Myocardial infarction, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting, New York Heart Association (NYHA) class III/IV congestive heart failure, cerebrovascular accident, transient ischemic attack, or rest leg claudication occurring within the 12 months prior to randomization;
8. Deep vein thrombosis or pulmonary embolism occurring within 6 months prior to randomization;
9. Any major surgery performed within 4 weeks prior to randomization;
10. A clear history of mental illness that hinders understanding of the informed consent and compliance with the study protocol;
11. Patients infected with the human immunodeficiency virus (HIV);
12. Active autoimmune diseases requiring systemic treatment in the past two years (such as treatment with disease-modifying drugs, corticosteroids, or immunosuppressants);
13. Subjects known to be allergic to similar drugs;
14. Any condition affecting the subject's ability to swallow medication or any condition affecting the absorption or pharmacokinetics of the investigational drug, including any history of gastrointestinal resection or surgery;
15. The presence of severe pulmonary disease, history of asthma or COPD, and pulmonary function tests indicating moderate to severe impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2028-12-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of initiate treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months until disease progression or death
  The definition of Progression-free survival（PFS） is the time from the date of first dose until the first observation of disease progression (PD) (as determined by radiographic assessment) or death (whichever occurs first).

SECONDARY OUTCOMES:
Overall survival | From date of initiate treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months until disease progression or death
  Overall survival（OS） was defined as the time from the date of first dose to the date of death from any cause.
Objective response rate | From date of initiate treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months until disease progression or death
  The Objective response rate（ORR） was defined as the proportion of patients with a best overall response of complete or partial response.
Disease control rate | From date of initiate treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months until disease progression or death
  Disease control rate（DCR）was defined the proportion of patients with complete response, partial response, and stable disease.
Duration of response | From date of initiate treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months until disease progression or death
  Duration of response (DOR)defined as the time from first documented response, PR or CR, to progressive disease [PD] or death; patients who neither progressed nor died were censored on the date of their last radiographic tumor assessment.
Dynamic changes in ctDNA levels and alterations in the ctDNA mutation profile | In this study, a maximum of six blood samples were collected for ctDNA testing, specifically before treatment, and after drug treatment at 2 months, 4 months, 6 months, 8 months, and at the time of PD (progressive disease) occurrence up to 36 months
  In this study, blood samples were collected for ctDNA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian F Zhou, M.D, Principal Investigator — 中山大学肿瘤防治中心
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No